CLINICAL TRIAL: NCT05323305
Title: Ultrasound Guided Pectointercostal Fascial Plane Block Versus Transversus Thoracic Plane Block In Adult Cardiac Surgery Patients: A Comparative Study
Brief Title: Pectointercostal Fascial Plane Block Versus Transversus Thoracic Plane Block In Adult Cardiac Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0305468
Record Dates: First submitted 2022-03-21; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Pain, Post Operative
Keywords: Ultrasound, pectointercostal, Cardiac surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pectointercostal Group (n=30) (Active Comparator): They will receive ultrasound-guided pectointercostal fascial block after induction of anesthesia with equal dose before extubation in the intensive care.
  Interventions: Procedure: ultrasound guided regional block
- Transversus thoracic Group (n=30) (Active Comparator): They will receive ultrasound-guided ultrasound-guided transversus thoracic plane block after induction of anesthesia with equal dose before extubation in the intensive care.
  Interventions: Procedure: ultrasound guided regional block

INTERVENTIONS:
Procedure: ultrasound guided regional block — Bupivacaine injection by the use of ultrasound in the pectointercostal fascial plane in one group and in the trasversus thoracic plane in the other group.
  Other Names: ultrasound guided nerve block

SUMMARY:
The study will be designed to compare the analgesic effect of ultrasound-guided pectointercostal fascial plane block versus tansversus thoracic plane block in adult cardiac surgery.

DETAILED DESCRIPTION:
A prospective study will be carried out in Alexandria Main University Hospitals on 60 adult patients planned for elective cardiac surgery, after approval of the Ethical Committee of Faculty of Medicine, Alexandria, and having an informed written consent taken from patients included in the study. Patients will be categorized into two equal groups; group P (n=30)) will receive ultrasound-guided pectointercostal fascial plane block and group T (n=30) will receive ultrasound-guided transversus thoracic plane block.

All patients will receive the ultrasound-guided block after induction of anesthesia and an equal booster dose of the same block before extubation in the ICU. Patients in both groups will also receive an ultrasound-guided bilateral serratus anterior plane block before extubation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient.
2. Elective cardiac surgery.

Exclusion Criteria:

1. Refusal to participate.
2. Redo or urgent cardiac surgery.
3. Local infection of the skin at the site of needle puncture.
4. Allergy to bupivacaine.
5. Coagulation disorders.
6. Clinically significant liver or kidney disease, heart failure, moderate to severe pulmonary hypertension.
7. when extubation is intentionally planned to be delayed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the analgesic effectiveness of the two blocks on midline sternotomy pain, | from end of surgery till discharge from ICU (96 hours)
  Postoperative pain evaluation after extubation will be done using the Visual Analogue Scale (VAS). a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 "no pain" and 10 "worst pain."

SECONDARY OUTCOMES:
pulmonary complications | from end of surgery till discharge from ICU (96 hours)
  atelectasis and pneumonia
length of stay in ICU | average 4 days
  days from admission till discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: islam Omar, MD, Study Chair — Lecturer of Anaesthesia and surgical intensive care, Faculty of medicine, Alexandria university; Ibrahim Ibrahim, MD, Principal Investigator — Lecturer of Anaesthesia and surgical intensive care, Faculty of medicine, Alexandria university; Moustafa Halwag, MD, Study Director — Lecturer of Anaesthesia and surgical intensive care, Faculty of medicine, Alexandria university
Locations (1):
- Alexandria University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately after publication No end date
Access Criteria: Any one who wishes to access the data